CLINICAL TRIAL: NCT02976402
Title: Stereotactic Hypofractionated Accelerated Radiotherapy Post-Prostatectomy: a Phase I Feasibility Study
Brief Title: Stereotactic Hypofractionated Accelerated Radiotherapy Post-Prostatectomy
Acronym: SHARP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Carlo Greco, MD, M.D., Fundacao Champalimaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARP
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer Adenocarcinoma; Adjuvant Radiotherapy; Salvage Radiotherapy; SBRT; IGRT; Urethral Sparing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT (Experimental): Postoperative RT consisting in:
  * 31 Gy in 5 sessions each of 6.2 Gy (adjuvant intent) delivered in one week
  * 32.5 Gy in 5 sessions each of 6.5 Gy (salvage intent) delivered in one week
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Postoperative RT consisting in:
  * 31 Gy in 5 sessions each of 6.2 Gy (adjuvant intent) delivered in one week
  * 32.5 Gy in 5 sessions each of 6.5 Gy (salvage intent) delivered in one week
  Other Names: Extremely Hypofractionationated Postoperative Radiotherapy for Prostate Cancer

SUMMARY:
The present phase I trial evaluates the feasibility of a postoperative stereotactic hypofractionated external beam radiation therapy delivered in patients who underwent radical prostatectomy with adverse pathological features or early biochemical failure. Modern computer-driven technology enables the implementation of ultra-high hypofractionated Image-Guided Radiotherapy (IGRT) safely.

Eligible patients for this study are those with:

* Adenocarcinoma of the prostate treated with radical prostatectomy (any type of radical prostatectomy is permitted including retropubic, perineal, laparoscopic or robotically assisted; there is no time limit for the date of radical prostatectomy)
* Pathologic (p)T3 disease, positive margin(s), Gleason score 8-10, or seminal vesicle involvement
* Undetectable post-radical prostatectomy PSA that becomes detectable and then increases on 2 subsequent measurements (PSA of > 0.1 - ≤ 2.0 ng/mL)
* Life expectancy: 10 years
* ECOG performance status of 0 -1
* No distant metastases, based on the following workup within 60 days prior to registration
* Magnetic resonance imaging (MRI) of the pelvis
* PSMA/Choline Positron Emission Tomography (PET) to exclude systemic disease in patients with biochemical recurrence
* Patients can be on androgen deprivation therapy
* Ability to understand and willingness to sign a study-specific informed consent prior to study.

Patients enrolled in the study will undergo image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility.

DETAILED DESCRIPTION:
The present study evaluates the feasibility of postoperative stereotactic hypofractionated external beam radiation therapy delivered in patients who underwent radical prostatectomy with adverse pathological features or early biochemical failure. Regardless the two settings (adjuvant or salvage), external beam radiation therapy for prostate cancer is usually a protracted course, since a total dose of 66 Gy to 70 Gy is needed to be effective. At the typical rate of 1.8 Gy to 2.0 Gy per treatment, it takes approximately 35 treatments over the course of 7 weeks to complete, which is very costly and extremely time consuming. On the other hand, the α/β ratio for prostate cancer has estimated to be as low as 1.5 Gy, significantly lower than the 3 Gy value estimated for late complications.Therefore, the delivery of the same equivalent total dose at 2 Gy/fraction (normalized total dose) to the prostate using a hypofractionation regimen, a part from the practical benefits of reducing the treatment cost and number of sessions for patients to radiotherapy departments, should have a sparing effect on early responding normal tissues through the reduction in the total dose delivered, as well as a reduction in the incidence of late complications. Trials investigating clinical and toxicity outcomes of moderate hypofractionation schedules in the curative setting have reached sufficient follow-up to show similar efficacy and toxicity to conventionally fractionated regimens.

Stereotactic body radiation therapy, or SBRT, is on the shortest end of the hypofractionation spectrum. It is accomplished in a five treatments. With its pinpoint accuracy, many Institutions currently use it for primary treatment at doses up to 9 Gy per treatment, leading to excellent outcomes at least at early time points.Patients enrolled in the study will undergo image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility.A rectal balloon with air filling will be used for anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients who underwent radical prostatectomy with adverse pathologic findings will be enrolled in a phase I study, consisting of 31 Gy (5 fractions of 6.2 Gy), respectively, delivered over a 1-week period at 5 fractions per week. This dosage corresponds to 68.2 Gy (for an α/βratio estimate of 1.5 Gy), compared to 52.7 Gy (for an α/β estimate of 4 Gy) in a conventional schedule. In those who developed early biochemical failure the radiation schedule will consists in 32.5 Gy (5 fractions of 6.5 Gy), respectively, delivered over a 1-week period at 5 fractions per week. This dosage corresponds to 74.3 Gy (for an α/β ratio estimate of 1.5 Gy), compared to 56.9 Gy (for an α/β estimate of 4 Gy) in a conventional schedule.

Patients will be followed at one month post-treatment and every 3 months for up to 12 months (+/- 4 weeks) and every 6 months thereafter. Acute and chronic toxicity evaluations will focus, though not exclusively, on urinary, rectal and sexual functions and will be assessed through validated EPIC questionnaires. Serum PSA values will be drawn on the same schedule as clinical follow-up. The study will be continuously monitored for a minimum of 5 years. In the event unexpected severe (grade ≥3) toxicities are observed in any one of the treatment regimens, the trial will be terminated according to the standard stopping rules: >3/first 10, and >5/first 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate treated with radical prostatectomy (any type of radical prostatectomy is permitted including retropubic, perineal, laparoscopic or robotically assisted; there is no time limit for the date of radical prostatectomy)
* Pathologic (p)T3 disease, positive margin(s), Gleason score 8-10, or seminal vesicle involvement
* Undetectable post-radical prostatectomy PSA that becomes detectable and then increases on 2 subsequent measurements (PSA of > 0.1 - ≤ 2.0 ng/mL)
* Life expectancy: 10 years
* ECOG performance status of 0 -1
* No distant metastases, based on the following workup within 60 days prior to registration
* Magnetic resonance imaging (MRI) of the pelvis
* PSMA/Choline Positron Emission Tomography (PET) to exclude systemic disease in patients with biochemical recurrence
* Patients can be on androgen deprivation therapy
* Ability to understand and willingness to sign a study-specific informed consent prior to study entry

Exclusion Criteria:

* N1 patients are ineligible, as are those with lymph node (LN) enlargement > 1.5 cm by computed tomography (CT) or MRI of the pelvis, unless the LN is biopsy proven to be negative.
* Gross residual disease in the prostate fossa based on imaging evidence, unless biopsy proven not to contain cancer.
* Prior radiation of any kind to the prostate gland or pelvis
* Prior brachytherapy is not allowed
* History of inflammatory colitis or other active severe comorbidities
* Patients who are on immunosuppressant medication

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility (ability to deliver radiation treatment as planned). | Participants should be followed continuously, for the duration of 5 years
  Monitoring treatment related adverse events as measured by Common Toxicity Criteria for Adverse Effects v4.0

SECONDARY OUTCOMES:
Number of participants with acute (≤ 90 days from treatment completion)treatment-related adverse events as assessed by CTCAE v4.0 | Participants should be followed continuously, for the duration of 5 years
Number of participants with late (> 90 days from treatment completion) treatment-related adverse events as assessed by CTCAE v4.0 with SBRT administered to the prostate bed | Participants should be followed continuously, for the duration of 5 years
Number of participants with post-treatment quality of life impairment assessed through validated tools (EPIC) | Participants should be followed continuously, for the duration of 5 years
Number of participants with post-treatment abnormal laboratory values (PSA relapse) | Participants should be followed continuously, for the duration of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, M.D., Principal Investigator — Champalimaud Foundation
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal